CLINICAL TRIAL: NCT03329196
Title: A Phase III, Open-label, Confirmatory Study of MT-6548 Compared to Darbepoetin Alfa in Non-dialysis Subjects With Anemia Associated With Chronic Kidney Disease in Japan
Brief Title: Efficacy and Safety Study to Evaluate MT-6548 in Non-dialysis Subjects With Anemia Associated With Chronic Kidney Disease in Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MT-6548-J01
Record Dates: First submitted 2017-10-30; First posted 2017-11-01 (Actual); Results first posted 2021-04-12 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Anemia; Non-dialysis Dependent Chronic Kidney Disease
MeSH Terms: conditions — Anemia | interventions — vadadustat; Darbepoetin alfa

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MT-6548 (Experimental)
  Interventions: Drug: MT-6548
- Darbepoetin alfa (Active Comparator)
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: MT-6548 — Oral tablet
  Other Names: vadadustat; AKB-6548
  Arms: MT-6548
Drug: Darbepoetin alfa — Subcutaneous
  Arms: Darbepoetin alfa

SUMMARY:
For Non-dialysis subjects with anemia associated with chronic kidney disease, demonstrate non-inferiority of MT-6548 compared to darbepoetin alfa using Hb value and evaluate long-term safety of MT-6548.

For subjects not currently receiving ESAs, evaluate Hb correction and maintenance effect of MT-6548 and for subjects currently receiving ESAs, evaluate Hb conversion and maintenance effect of MT-6548

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CKD
* eGFR < 60 mL/min/1.73m^2 during the screening period
* Not receiving dialysis for 8 weeks prior to the screening period, and not expected to start dialysis during the treatment period
* Correction group: Not being treated with ESAs for the recent 8 weeks prior to the screening period
* Conversion group: Being treated with ESAs for the recent 8 weeks prior to the screening period
* Mean of the two screening Hb levels closest in time to the baseline visit. Correction group: ≥8.0 g/dL and < 11.0 g/dL Conversion group: ≥9.0 g/dL and ≤12.5 g/dL
* Fluctuation between the two Hb levels closest in time to the baseline visit during the screening period less than 1.5 g/dL
* Serum ferritin ≥ 100 ng/mL, or TSAT ≥20% during the screening period
* Folate and vitamin B12 ≥ lower limit of normal during the screening period

Exclusion Criteria:

* Anemia due to a main cause other than CKD: sickle cell disease, myelodysplastic syndrome, bone marrow fibrosis, hematologic malignancy, hemolytic anemia, thalassemia, or pure red cell aplasia
* Active bleeding or recent blood loss within 8 weeks prior to the screening period
* RBC transfusion within 8 weeks prior to the screening period
* Received testosterone enanthate or mepitiostane within 8 weeks prior to the screening period
* AST, ALT, or total bilirubin >2.5 x upper limit of normal during the screening period
* Uncontrolled hypertension (diastolic blood pressure >110 mm Hg or systolic blood pressure >180 mm Hg) during the screening period and Day 1
* Ophthalmic examinations during the screening period correspond to either of the following criteria;

  * No available fundal findings
  * Findings indicating the presence of active fundal disease
* Severe heart failure (New York Heart Association Class IV)
* Cerebrovascular disorder or acute coronary syndrome (hospitalization due to unstable angina or myocardial infarction), requiring hospitalization due to urgent percutaneous intervention for coronary or heart failure within 12 weeks prior to the screening period
* Current or history of malignancy. History of malignancy with no recurrence for the recent 5 years is not an exclusion criterion
* New onset or recurrent event of deep vein thrombosis or pulmonary embolism within 12 weeks prior to the screening period
* Current or history of hemosiderosis or hemochromatosis
* History of prior organ transplantation or scheduled organ transplant, or prior transplantation of hematopoietic stem cell or bone marrow
* Males and females of childbearing potential who are unwilling to use an acceptable method of contraception during the designated period (Males: during the study and 90 days after the last dose, females: during study and 30 days after the last dose)
* Females who are pregnant or breast feeding, or are predicted to be pregnant

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (31):
- Japan (31):
  - Research site, Aichi
  - Research site, Chiba
  - Research site, Fukui
  - Research site, Fukuoka
  - Research site, Fukushima
  - Research site, Gunma
  - Research site, Hiroshima
  - Research site, Hokkaido
  - Research site, Hyōgo
  - Research site, Ibaraki
  - Research site, Kagoshima
  - Research site, Kanagawa
  - Research site, Kochi
  - Research site, Kumamoto
  - Research site, Kyoto
  - Research site, Miyagi
  - Research site, Nagano
  - Research site, Nagasaki
  - Research site, Nara
  - Research site, Niigata
  - Research site, Okayama
  - Research site, Okinawa
  - Research site, Osaka
  - Research site, Ōita
  - Research site, Saga
  - Research site, Saitama
  - Research site, Shiga
  - Research site, Shizuoka
  - Research site, Tokyo
  - Research site, Toyama
  - Research site, Yamanashi

REFERENCES:
- [Result] Nangaku M, Kondo K, Kokado Y, Ueta K, Kaneko G, Tandai T, Kawaguchi Y, Komatsu Y. Phase 3 Randomized Study Comparing Vadadustat with Darbepoetin Alfa for Anemia in Japanese Patients with Nondialysis-Dependent CKD. J Am Soc Nephrol. 2021 Jul;32(7):1779-1790. doi: 10.1681/ASN.2020091311. Epub 2021 Apr 21. PMID 33883252
- [Derived] Nangaku M, Ueta K, Nishimura K, Sasaki K, Hashimoto T. Factors affecting responsiveness of vadadustat in patients with anemia associated with chronic kidney disease: a post-hoc subgroup analysis of Japanese phase 3 randomized studies. Clin Exp Nephrol. 2024 May;28(5):391-403. doi: 10.1007/s10157-023-02432-z. Epub 2024 Mar 26. PMID 38530490
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278

RESULTS

PARTICIPANT FLOW:
Groups:
- MT-6548: MT-6548: Oral tablet. The dose was adjusted to 150-600 mg/day according to the pre-specified dose adjustment algorithm.
- Darbepoetin Alfa: Darbepoetin alfa: Subcutaneous. The dose was adjusted to 15-180 ug/week, 2 weeks or 4 weeks according to the pre-specified dose adjustment algorithm.
Period: Overall Study
Arm/Group | MT-6548 | Darbepoetin Alfa
Started | 151 | 153
Completed | 111 | 123
Not Completed | 40 | 30
Not completed — Adverse Event | 10 | 5
Not completed — Physician Decision | 2 | 2
Not completed — Withdrawal by Subject | 11 | 3
Not completed — Hepatic function abnormalities | 0 | 1
Not completed — Conducting rescue therapy before Week 24 | 2 | 1
Not completed — Difficult to control Hb | 2 | 3
Not completed — Dialysis or renal transplant | 13 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MT-6548 | Darbepoetin Alfa | Total
Number analyzed (Participants) | 151 | 153 | 304
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 28 | 61
  >=65 years | 118 | 125 | 243
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 80 | 156
  Male | 75 | 73 | 148
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian (Japanese) | 151 | 153 | 304
  Asian (Other) | 0 | 0 | 0
  Other | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Hb Level of Week 20 and Week 24
Time Frame: Up to Week 24
Measure: Least Squares Mean (95% Confidence Interval); unit: g/dL
Arm/Group | MT-6548 | Darbepoetin Alfa
Number analyzed (Participants) | 151 | 153
g/dL | 11.66 [11.49 to 11.84] | 11.93 [11.76 to 12.10]

2. Secondary Outcome: Mean Hb Level of Week 48 and Week 52
Time Frame: Up to Week 52
Measure: Least Squares Mean (95% Confidence Interval); unit: g/dL
Arm/Group | MT-6548 | Darbepoetin Alfa
Number analyzed (Participants) | 151 | 153
g/dL | 11.54 [11.38 to 11.69] | 11.63 [11.48 to 11.77]

3. Secondary Outcome: Hb Level at Each Assessment Time Point
Time Frame: Up to Week 52
Population: This analysis was performed only in subjects who have Hb data at each visit.
Measure: Mean (95% Confidence Interval); unit: g/dL
Arm/Group | MT-6548 | Darbepoetin Alfa
Number analyzed (Participants) | 151 | 153
g/dL
  Baseline | 10.44 [10.29 to 10.59] | 10.52 [10.38 to 10.66]
  Week 2 | 10.64 [10.48 to 10.80] | 10.75 [10.62 to 10.89]
  Week 4: number analyzed (Participants) | 149 | 152
  Week 4 | 10.71 [10.54 to 10.89] | 10.90 [10.76 to 11.05]
  Week 6: number analyzed (Participants) | 148 | 152
  Week 6 | 10.87 [10.69 to 11.04] | 11.23 [11.08 to 11.38]
  Week 8: number analyzed (Participants) | 145 | 151
  Week 8 | 11.13 [10.96 to 11.30] | 11.42 [11.26 to 11.59]
  Week 10: number analyzed (Participants) | 145 | 150
  Week 10 | 11.33 [11.17 to 11.49] | 11.70 [11.54 to 11.85]
  Week 12: number analyzed (Participants) | 145 | 148
  Week 12 | 11.50 [11.34 to 11.67] | 11.88 [11.72 to 12.04]
  Week 16: number analyzed (Participants) | 143 | 148
  Week 16 | 11.56 [11.39 to 11.74] | 12.00 [11.84 to 12.16]
  Week 20: number analyzed (Participants) | 139 | 144
  Week 20 | 11.66 [11.47 to 11.84] | 11.92 [11.77 to 12.06]
  Week 24: number analyzed (Participants) | 132 | 140
  Week 24 | 11.68 [11.49 to 11.87] | 11.94 [11.80 to 12.08]
  Week 28: number analyzed (Participants) | 125 | 137
  Week 28 | 11.72 [11.56 to 11.88] | 11.89 [11.74 to 12.03]
  Week 32: number analyzed (Participants) | 120 | 132
  Week 32 | 11.74 [11.57 to 11.91] | 11.79 [11.66 to 11.92]
  Week 36: number analyzed (Participants) | 119 | 129
  Week 36 | 11.74 [11.58 to 11.91] | 11.99 [11.84 to 12.15]
  Week 40: number analyzed (Participants) | 114 | 127
  Week 40 | 11.61 [11.46 to 11.76] | 11.78 [11.66 to 11.91]
  Week 44: number analyzed (Participants) | 114 | 124
  Week 44 | 11.50 [11.35 to 11.66] | 11.68 [11.56 to 11.80]
  Week 48: number analyzed (Participants) | 110 | 124
  Week 48 | 11.68 [11.52 to 11.84] | 11.73 [11.59 to 11.87]
  Week 52: number analyzed (Participants) | 109 | 122
  Week 52 | 11.62 [11.47 to 11.77] | 11.64 [11.52 to 11.76]
  Week 52 (LOCF) | 11.29 [11.11 to 11.47] | 11.50 [11.34 to 11.65]

4. Secondary Outcome: Percentage of Subjects With Hb Level at Each Assessment Time Point Within the Target Range During the Treatment Period
Time Frame: Up to Week 52
Population: This analysis was performed only in subjects who have Hb data at each visit.
Measure: Number; unit: percentage of subjects
Arm/Group | MT-6548 | Darbepoetin Alfa
Number analyzed (Participants) | 151 | 153
percentage of subjects
  Baseline | 31.1 | 32.7
  Week 2 | 36.4 | 37.9
  Week 4: number analyzed (Participants) | 149 | 152
  Week 4 | 46.3 | 53.3
  Week 6: number analyzed (Participants) | 148 | 152
  Week 6 | 45.3 | 63.8
  Week 8: number analyzed (Participants) | 145 | 151
  Week 8 | 57.9 | 65.6
  Week 10: number analyzed (Participants) | 145 | 150
  Week 10 | 59.3 | 68.0
  Week 12: number analyzed (Participants) | 145 | 148
  Week 12 | 68.3 | 67.6
  Week 16: number analyzed (Participants) | 143 | 148
  Week 16 | 68.5 | 71.6
  Week 20: number analyzed (Participants) | 139 | 144
  Week 20 | 65.5 | 73.6
  Week 24: number analyzed (Participants) | 132 | 140
  Week 24 | 68.2 | 77.9
  Week 28: number analyzed (Participants) | 125 | 137
  Week 28 | 77.6 | 76.6
  Week 32: number analyzed (Participants) | 120 | 132
  Week 32 | 75.0 | 78.8
  Week 36: number analyzed (Participants) | 119 | 129
  Week 36 | 77.3 | 77.5
  Week 40: number analyzed (Participants) | 114 | 127
  Week 40 | 76.3 | 87.4
  Week 44: number analyzed (Participants) | 114 | 124
  Week 44 | 71.9 | 85.5
  Week 48: number analyzed (Participants) | 110 | 124
  Week 48 | 74.5 | 79.8
  Week 52: number analyzed (Participants) | 109 | 122
  Week 52 | 75.2 | 80.3

5. Secondary Outcome: Time to Reach the Target Hb Range in Correction Group Only
Time Frame: Up to Week 52
Population: This analysis was performed in correction group except for subjects with Hb is 11.0 g/dL or more at baseline.
Measure: Median (Full Range); unit: days
Arm/Group | MT-6548 | Darbepoetin Alfa
Number analyzed (Participants) | 60 | 64
days | 43.0 [12 to 361] | 29.0 [14 to 225]

6. Secondary Outcome: Rate of Increase in Hb Level in Correction Group Only
Time Frame: Up to Week 6
Population: This analysis was performed in subjects of correction group who have Hb up to week 4 or week 6.
Measure: Mean (95% Confidence Interval); unit: g/dL/week
Arm/Group | MT-6548 | Darbepoetin Alfa
Number analyzed (Participants) | 69 | 70
g/dL/week
  Calculated based on Hb at baseline and Week 4 | 0.14 [0.09 to 0.19] | 0.21 [0.17 to 0.24]
  Calculated based on Hb up to Week6 | 0.13 [0.09 to 0.17] | 0.21 [0.18 to 0.25]

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | MT-6548 | Darbepoetin Alfa
All-Cause Mortality (participants affected / at risk) | 0/151 | 1/153
Serious Adverse Events (participants affected / at risk) | 42/151 | 49/153
Other Adverse Events (participants affected / at risk) | 85/151 | 80/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MT-6548 (N=151) | Darbepoetin Alfa (N=153)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 2
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Cataract (Eye disorders) | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 2
Ischaemic enteritis (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 1
Oesophageal achalasia (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 2
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 1
Mediastinal abscess (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Periodontitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 3
Pneumonia chlamydial (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Renal cyst infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Shunt occlusion (Injury, poisoning and procedural complications) | 0 | 1
Shunt stenosis (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypoglycaemic coma (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 7 | 11
Diabetic nephropathy (Renal and urinary disorders) | 0 | 1
End stage renal disease (Renal and urinary disorders) | 3 | 1
Renal failure (Renal and urinary disorders) | 2 | 1
Renal impairment (Renal and urinary disorders) | 6 | 6
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 | 0
Peripheral artery aneurysm (Vascular disorders) | 0 | 1
Vascular rupture (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MT-6548 (N=151) | Darbepoetin Alfa (N=153)
Constipation (Gastrointestinal disorders) | 14 | 11
Diarrhoea (Gastrointestinal disorders) | 18 | 8
Vomiting (Gastrointestinal disorders) | 10 | 3
Oedema peripheral (General disorders) | 11 | 5
Pyrexia (General disorders) | 8 | 1
Cystitis (Infections and infestations) | 6 | 9
Nasopharyngitis (Infections and infestations) | 37 | 43
Contusion (Injury, poisoning and procedural complications) | 11 | 7
Chronic kidney disease (Renal and urinary disorders) | 5 | 8
Eczema (Skin and subcutaneous tissue disorders) | 5 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 8
Hypertension (Vascular disorders) | 2 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/96/NCT03329196/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-06): https://cdn.clinicaltrials.gov/large-docs/96/NCT03329196/SAP_001.pdf